CLINICAL TRIAL: NCT03651726
Title: A Randomized Double Blind Placebo Controlled Proof of Concept Study to Evaluate Safety, Tolerability and Efficacy of Daily Oral THX-110 in Treating Adults With Tourette Syndrome ("Entourage")
Brief Title: A Study to Examine the Efficacy of a Therapeutic THX-110 for Tourette Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Neurothera Labs Inc. (Industry)
Collaborators: FGK Clinical Research GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: THX-G18-001
Record Dates: First submitted 2018-08-09; First posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Tourette Syndrome
MeSH Terms: conditions — Tourette Syndrome | interventions — Dronabinol; palmidrol

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo controlled, proof of concept study, followed by an open uncontrolled treatment phase
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- THX-110 (dronabinol plus PEA) (Experimental): Double-blind phase and extension open label phase:
  Dose range of 2.5 mg to 10 mg dronabinol (1 to 4 capsules) plus 800 mg PEA (2 tablets) taken orally once daily; starting dose is 2.5 mg dronabinol plus 800 mg PEA. Up-titration is performed within maximal 3 weeks. The titration phase is followed by a maintenance phase of 9 weeks at stable dose.
  Interventions: Drug: THX-110 (dronabinol plus PEA)
- Placebo (Placebo Comparator): Double-blind phase:
  Range of 1 to 4 dronabinol placebo capsules plus 2 PEA placebo tablets taken orally once daily; starting dose is 1 dronabinol placebo capsule plus 2 PEA placebo tablets. Up-titration is performed within maximal 3 weeks. The titration phase is followed by a maintenance phase of 9 weeks at stable dose.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: THX-110 (dronabinol plus PEA) — 2.5 mg dronabinol capsules and 400 mg PEA tablets
  Other Names: Dronabinol; Tetrahydrocannabinol; THC; Palmidrol; Palmitoylethanolamide
  Arms: THX-110 (dronabinol plus PEA)
Drug: Placebo — Sesame oil pill manufactured to mimic 2.5 mg dronabinol capsules; cellulose pill manufactured to mimic 400 mg PEA tablets
  Arms: Placebo

SUMMARY:
This study evaluates the efficacy and safety of THX-110 in the management of tics and other symptoms (e.g. rage attacks, anxiety, depression, sleep difficulties) in patients with Tourette syndrome. In the first part of the study, half of the patients will receive THX-110, while the other half will receive a placebo. After completion of the first study part, patients will have the opportunity to continue into the second part of the study. In this part, all participants will receive THX-110.

DETAILED DESCRIPTION:
THX-110 is an investigational drug and is being developed for the treatment of patients with Tourette syndrome and other conditions. THX-110 consists of an active substance from cannabis (dronabinol, tetrahydrocannabinol, THC) and PEA, a substance that occurs naturally in the human body, in animals and plants.

Dronabinol and similar active substances are already approved in some countries for the treatment of other conditions. In some countries, various cannabis-based medications are currently being used in the treatment of patients with Tourette syndrome, mostly without official approval.

PEA has already been used and well tolerated in numerous clinical trials. The combination of PEA and dronabinol is assumed to show better efficacy compared to treatment with dronabinol alone.

The planned study will evaluate the efficacy of THX-110 in the management of tics and other symptoms in patients with Tourette syndrome. Other objectives are to assess study drug dosage and to identify side effects that may be associated with the study drug.

In the first part of the study, half of the patients will receive THX-110, while the other half will receive a placebo. The treatment phase will last 12 weeks. After completion of the first part, patients can decide if they want to participate in the second part of the study. In this optional second part of the study, all patients will receive THX-110 for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Tourette syndrome according to DSM-5
2. Male and female subjects with an age between ≥18 and <65 years
3. Total tic score (TTS) of the YGTSS >18
4. CGI-S ≥4
5. Medication (and stimulation parameters for deep brain stimulation) for tics and comorbidities must be on a stable dose for at least 6 weeks before entering the study and subject must consent to maintain the stable dose during the study
6. Signed written informed consent and willingness to comply with treatment and follow-up procedures
7. Subjects capable of understanding the investigational nature, potential risks and benefits of the clinical study
8. Women of child-bearing potential must have a negative pregnancy test (i.e., negative for urine human chorionic gonadotropin [hCG]) before first treatment with study medication. They must practice a highly effective, reliable and medically approved contraceptive regimen during the study (e.g., theoretical failure rate less than 1% per year a when used consistently and correctly), which include oral or parenteral or implanted hormonal contraception, vaginal ring releasing hormonal contraception (e.g., Nuvaring), intrauterine device or intrauterine system. Post-menopausal women may enter this study. Post-menopausal women are defined as those without menses in the past 12 months without an alternative medical cause, and with a serum follicle stimulating hormone (FSH) in the post-menopausal range. Women who are surgically sterile may enter this study with historical documentation of surgical procedure (bilateral tubal ligation or bilateral oophorectomy at least 6 weeks prior screening or hysterectomy or uterine agenesis) and a negative pregnancy test.
9. Male subjects must be willing to use a condom with sexual partners during this study and for a period of three months following the last administration of study medication until the follow-up visit. Male subjects must be willing to abstain from sperm donation for 3 months after the completion of this study.

Exclusion Criteria:

1. Comorbid OCD, ADHD, depression, or anxiety disorder when unstable and/or in need of an initial adjustment for a therapy
2. Presence of a comorbid psychiatric condition as developmental disability, psychotic illness or bipolar disorder
3. Ongoing behavioural treatment for tics
4. History of schizophrenia, seizure, psychotic, severe personality, or pervasive developmental disorder
5. Current clinical diagnosis of substance abuse or dependence
6. History of cannabis dependence
7. Secondary and other chronic tic disorders or other significant neurological disorders
8. History of severe cardiac diseases, severe cardiovascular diseases, severe renal disorders, or severe hepatic diseases and/or positive for human immunodeficiency virus (HIV), hepatitis C, or hepatitis B
9. Concomitant medications have to be on stable dose since at least 6 weeks before entering the study and must be well tolerated at baseline without causing dizziness, confusion, sedation, or somnolence such as central nervous system depressants (e.g., barbiturates, benzodiazepines, ethanol, lithium, opioids, buspirone, scopolamine, antihistamines, tricyclic antidepressants, other anticholinergic agents, muscle relaxants)
10. Use of cannabis or CBM in the 30-day period prior to study entry and/or positive delta-9-THC urine test at baseline
11. Positive pregnancy test, i.e., positive for urine beta-hCG
12. Pregnant or breast-feeding women
13. Subjects who received any investigational medication or used any investigational device within 30 days prior to the first dose of study medication or is actively participating in any investigational drug or device study, or is scheduled to receive an investigational drug or to use an investigational device during the course of the study
14. Subjects with a known allergy, hypersensitivity, or intolerance to the active substances and/or excipients of study medication (e.g., cannabis, cannabinoids, sesame oil)
15. Any condition, which in the opinion of the investigator, would interfere with the evaluation of the study product or poses a health risk to the subject
16. Subjects who are employees of the sponsor or employees or close relatives of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-11 (Estimated); Study Completion 2019-11 (Estimated)

PRIMARY OUTCOMES:
Change in YGTSS-TTS | Baseline and week 12 of the double-blind phase
  Absolute change in YGTSS-TTS as a continuous endpoint at week 12 of the double-blind phase (visit 9) compared to baseline.

SECONDARY OUTCOMES:
Response to treatment according to YGTSS-TTS | Baseline and week 12 of the double-blind phase
  Key secondary endpoint is the response to treatment according to YGTSS-TTS, defined as a reduction in YGTSS-TTS of at least 20% (compared to baseline) at week 12 of the double-blind phase (visit 9).
YGTSS-TTS as a binary responder criterion and as a continuous endpoint at week 7 of the double-blind phase | Baseline and week 7 of the double-blind phase
YGTSS-GS (= YGTSS-TTS + YGTSS-impairment score) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
Modified Rush Video-Based Tic Rating Scale (MRVS) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  No. of Body Areas (score 0-4), Motor Tic Frequency (tics/min) (score 0-4) Phonic Tic Frequency (score 0-4) Severity of Motor Tics (score 0-4) Severity of Phonic Tics (score 0-4) Total score (0-20) 0=best, 20=worst
Clinical Global Impression-Improvement Score (CGI-I) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The CGI-S score obtained at the baseline (initiation) visit serves as a good basis for making this assessment. Only the following one query is rated on a seven-point scale: "Compared to the patient's condition at admission to the project [prior to medication initiation], this patient's condition is: 1=very much improved since the initiation of treatment; 2=much improved; 3=minimally improved; 4=no change from baseline (the initiation of treatment); 5=minimally worse; 6= much worse; 7=very much worse since the initiation of treatment."
Clinical Global Impression-Severity Score (CGI-S) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The CGI-Severity (CGI-S) asks the clinician one question: "Considering your total clinical experience with this particular population, how mentally ill is the patient at this time?" which is rated on the following seven-point scale: 1=normal, not at all ill; 2=borderline mentally ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill patients.
  This rating is based upon observed and reported symptoms, behavior, and function in the past seven days. Clearly, symptoms and behavior can fluctuate over a week; the score should reflect the average severity level across the seven days.
Adult Tic Questionnaire (ATQ) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The ATQ includes a list of 14 common motor tics and 131 common vocal tics. For each type of tic, participants are asked to indicate its presence during the past week by selecting "yes" or "no." Subsequently, for each tic endorsed, participants indicate its frequency and intensity, both on a 4-point Likert-type scale. For the frequency ratings, scores range from a few times a week or less (1), to constantly, almost all the time during the day (4). For the intensity ratings, participants are asked to check (1) if the specific tic was very mild in intensity in the past week, (2) or higher if the tic was obviously noticeable to others; and 3 or higher if the tic was much more forceful and very noticeable to others during the past week. A separate score of tic severity was calculated by summing the intensity and frequency score, resulting in a score between 2 (minimal frequency and intensity) to 8 (maximum frequency and intensity) for each tic endorsed.
Tourette Syndrome-Quality of Life Scale (GTS-QoL) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  HRQOL is often measured by four core questions that asked about general health status and number of unhealthy days in the Behavioral Risk Factor Surveillance System (BRFSS).
  HrQoL in GTS patients is evaluated using the generic EQ-5D instrument (ref: EuroQol-Group. EQ-5D. Available at:www.euroqol.org. 2006.). It includes a five dimension descriptive system and a visual analog scale (EQVAS). The five dimensions include ''Mobility,'' ''Self-Care,'' ''Usual Activities,'' ''Pain/Discomfort,'' and ''Anxiety/Depression.'' All dimensions are subdivided into three levels (no problems, some problems, and extreme problems). Calculation of EQ-5D index score was performed using a regression algorithm generated by Greiner et al (ref: Greiner W, et al. The measurement and valuation of health status using EQ-5D: a European perspective. Dordrecht: Kluwer Academic Publisher; 2003.)
Pre-monitory Urge for Tics Scale (PUTS) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The PUTS is a 9-item self-report questionnaire measuring premonitory sensations in individuals with tics. Each item is scored from 1 (not at all true) to 4 (very much true). The total score is computed by summing the 9 items. Thus, total scores range from 9 to 36, and higher scores represent greater premonitory urges. The PUTS has demonstrated good internal consistency, test-retest reliability, and construct validity among youths between 11 and 16 years of age.The present manuscript reports the first psychometric data on the 9-item PUTS in an older adolescent and adult sample.
Beck Depression Inventory (BDI) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  Add up the score for each of the twenty-one questions. The highest possible total for the whole test would be sixty-three. This would mean the number three was answered on all twenty-one questions. Since the lowest possible score for each question is zero, the lowest possible score for the test would be zero.
  Total Score____________________Levels of Depression 1-10____________________These ups and downs are considered normal 11-16___________________ Mild mood disturbance 17-20___________________Borderline clinical depression 21-30___________________Moderate depression 31-40___________________Severe depression over 40__________________Extreme depression
Yale-Brown Obsessive Compulsive Scale (Y BOCS) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The YBOCS is a 10-item clinician-rated measure of OCD symptom severity. Raters assess obsessions and compulsions separately in five domains: time spent, interference, distress, resistance, and control. Each domain is rated on a scale from 0 to 4. Thus, total scores range from 0 to 40, with higher scores indicating greater symptom severity.
Conners' Adult ADHD Rating Scale (CAARS) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The self-report and observer forms contain an identical set of scales, subscales, and indexes with a total of 30 items : Total ADHD symptoms: Inattentive (9 items), Hyperactive-Impulsive (9 items) subscales and ADHD Index (12 items) with each item rated on a 4-point scale (0=never, 1= a little, 2=often, 3= frequently) derived from from Conners' ADHD Rating Scale (CARS).
Beck Anxiety Inventory (BAI) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The total score is calculated by finding the sum of the 21 items. Score of 0-21 = low anxiety Score of 22-35 = moderate anxiety Score of 36 and above = potentially concerning levels of anxiety
Pittsburgh Sleep Quality Index (PSQI) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The Pittsburgh Sleep Quality Index (PSQI) contains 19 self-rated questions and 5 questions rated by the bed partner or roommate (if one is available). Only self-rated questions are included in the scoring. The 19 self-rated items are combined to form seven "component" scores, each of which has a range of 0-3 points. In all cases, a score of "0" indicates no difficulty, while a score of "3" indicates severe difficulty. The seven component scores are then added to yield one "global" score, with a range of 0-21 points, "0" indicating no difficulty and "21 " indicating severe difficulties in all areas.
12-item short-form (SF-12) Health Survey | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase
  The SF-12 is a multipurpose short form survey with 12 questions, all selected from the SF-36 Health Survey. The questions were combined, scored, and weighted to create two scales that provide glimpses into mental and physical functioning and overall health-related-quality of life.
  Physical and Mental Health Composite Scores (PCS & MCS) are computed using the scores of twelve questions and range from 0 to 100, where a zero score indicates the lowest level of health measured by the scales and 100 indicates the highest level of health.
Rage Attacks Questionnaire (RAQ) | Baseline, week 7 and week 12 of the double-blind phase, week 19 and week 24 of the extension open label phase

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Müller-Vahl, Prof. Dr., Study Chair — Medizinische Hochschule Hannover, Klinik für Psychiatrie, Sozialpsychiatrie und Psychotherapie
Locations (2):
- Germany (2):
  - Medizinische Hochschule Hannover, Klinik für Psychiatrie, Sozialpsychiatrie und Psychotherapie, Hanover
  - LMU Klinikum der Universität München, Klinik für Psychiatrie und Psychotherapie, Munich

IPD SHARING:
Plan to Share IPD: Undecided